CLINICAL TRIAL: NCT07168759
Title: An Educational Intervention Using a Virtual Reality Game to Improve Compliance With Coronavirus 2019 Disease-related Hygiene Practices and Participation in Severe Acute Respiratory Syndrome Virus 2 (SARS-CoV-2) Screening, for the Prevention of SARS-CoV-2 Transmission Between Primary Schoolchildren in Communities: a Stratified Cluster-randomised Controlled Trial
Brief Title: Educational VR Game Intervention to Enhance Hygiene Practices in Primary School Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMRF2025
Record Dates: First submitted 2025-07-17; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: VR games; Hygiene compliance; Hand hygiene; Upper respiratory tract infections; Schoolchildren
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): School children will participate in a VR game-based education programme
  Interventions: Other: VR game -based education program
- Control group (No Intervention): Schoolchildren in this group will receive the usual health education

INTERVENTIONS:
Other: VR game -based education program — The schoolchildren in the intervention group participate in an innovative VR game-based educational programme featuring: (1) Web-based health education on (i) SARS-CoV-2 and Influenza virus transmission, (ii) proper hand and respiratory hygiene practices and (iii) the importance of rapid screening and vaccination in the prevention of upper respiratory tract infections.
  Arms: Intervention group

SUMMARY:
The goal of this observational study is to investigate if VR game-based educational intervention can enhance primary schoolchildren's compliance with hygiene practices to prevent the transmission of SARS-CoV-2 and other upper respiratory pathogens in the community.

The main questions the study aims to answer are, after receiving the VR game-based education intervention:

* Does VR game-based educational intervention improve hygiene-practice compliance in primary schoolchildren?
* What are the bacterial loads on primary schoolchildren's hands?
* What are the rates of infections caused by SARS-CoV-2 and other respiratory viruses in primary schoolchildren?

Researchers will compare the interventional group to the control group to see if VR game-based educational intervention can enhance primary schoolchildren's hygiene practices.

Participants will

* Receive in a training programme on hygiene practices through playing VR games for two weeks, 1 hour per week.
* Do a questionnaire on hygiene knowledge before and after receiving the education programme
* Provide hand swabs and saliva samples before and after receiving the education programme

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a VR game (VRG)-based educational program on hygiene practices among primary schoolchildren in Hong Kong. The research design employs a randomized controlled trial with repeated measures.

Participants will be primary schoolchildren aged 6 to 12 who can communicate and read in Chinese. To minimize selection bias, children will remain unaware of their group assignments. The sample size calculation aims for a statistical power of at least 0.8, targeting 2160 participants across 18 school clusters. Thirty-six local primary schools will be randomly assign to the intervention group or the control group in a ratio of 1:1.

The pilot phase will refine the VRG educational program based on feedback from a previous intervention. Two schools will be selected for this pilot, where trained teachers will assist in student recruitment. The main intervention will involve an VRG-based educational program delivered over two to three weeks. Children in the intervention group will engage with VRGs that cover topics such as SARS-CoV-2 and influenza virus transmission, hygiene practices, importance of rapid testing and vaccination in the prevention of upper respiratory tract infections. The control group will receive standard community health education and will be invited to participate in the VRG program after the intervention period.

Each child's involvement will last six months, with assessments occurring at baseline (T1) and at two subsequent intervals: immediately-post (T2), 1-month post (T3). Data collection will include demographic data, questionnaire to assesses hygiene knowledge, videos to record handwashing practices, hand swabs to measures bacterial loads on hands and saliva samples to tests for respiratory viruses.

ELIGIBILITY:
Inclusion Criteria:

* Primary schoolchildren aged 6-12 years.
* Able to communicate in Chinese and to read Chinese.

Exclusion Criteria:

* Reported mental or physical health disorders.
* Participated in other health educational programs related to hygiene practices 2 months or less before recruitment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2160 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the compliance with hygiene practices immediately after intervention | Day 0, Month 1, Month 2
  Knowledge of hygiene practices assessed through a true/false questionnaire.
Change from baseline in the number of participants who comply with hand washing procedures immediately after intervention | Day 0, Month 1, Month 2
  Hand washing procedure compliance measured using video recordings.
Change from baseline in the number of bacteria on the hands of the participants immediately after intervention | Day 0, Month 1, Month 2
  Bacterial counts on the hands of participants will be assessed using hand swab sampling and quantitative microbiological analysis. Specifically, hand swabs will be collected from the participants before and after intervention. This will be followed by using plate count method to detect the number of bacterial cells present on the hand swabs collected from the participants.
Change from baseline in the vaccination uptake rates by the participants immediately after intervention | Day 0, Month 1, Month 2
  Data on vaccination uptake rates will be collected from the participants using a standardized questionnaire before and after intervention. The data will be aggregated to calculate the percentage change in vaccination uptake rates from pre- to post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No